CLINICAL TRIAL: NCT02664350
Title: Precision Medicine Guided Treatment for Cancer Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB201500780; OCR16264 (Other: University of Florida)
Record Dates: First submitted 2016-01-22; First posted 2016-01-27 (Estimated); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Pain; CYP2D6 Polymorphism
MeSH Terms: conditions — Pain | interventions — Cytochrome P-450 CYP2D6

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Genotype Arm (Experimental): Participants in this arm will have genotyping performed for CYP2D6 variants. Based on the CYP2D6 the treating physicians will be provided with an interpretation of genotype results, and a recommendation will be provided by a pharmacist on the UF Health Personalized Medicine team through one-on-one consultation with the physician for the type of pain medication. These participants will also be genotyped for OPRM1 variants at the end of the study which is performed for research purposes only. In addition, they will fill out the following questionnaires Brief Pain Inventory-Short Form (BPI-SF) and M.D. Anderson Symptom Inventory (MDASI).
  Interventions: Genetic: CYP2D6; Behavioral: Brief Pain Inventory-Short Form (BPI-SF); Behavioral: M.D. Anderson Symptom Inventory (MDASI); Genetic: OPRM1
- Traditional Arm (Active Comparator): Participants in this arm will have genotyping for CYP2D6 and OPRM1, however this information will not be provided to the physicians for treatment of the analgesic therapy but will be used for research purposes only. In addition, they will fill out the following questionnaires Brief Pain Inventory-Short Form (BPI-SF) and M.D. Anderson Symptom Inventory (MDASI).
  Interventions: Genetic: CYP2D6; Behavioral: Brief Pain Inventory-Short Form (BPI-SF); Behavioral: M.D. Anderson Symptom Inventory (MDASI); Genetic: OPRM1

INTERVENTIONS:
Genetic: CYP2D6 — Gentic testing for CYP2D6 metabolic pathway will be performed at baseline.
  Other Names: cytochrome P450 2D6
Behavioral: Brief Pain Inventory-Short Form (BPI-SF) — This questionnaire will be completed at baseline and weeks 2, 4, 6 and 8.
Behavioral: M.D. Anderson Symptom Inventory (MDASI) — This questionnaire will be completed at baseline and weeks 2, 4, 6 and 8.
Genetic: OPRM1 — Genetic testing of the OPRM1 will be performed after week 8.
  Other Names: µ-opioid receptor gene

SUMMARY:
Pain is one of the most burdensome symptoms associated with cancer and its treatment, and opioids are the cornerstone of clinical pain management in cancer patients. Yet, individual patient responses to opioids vary widely, and the patient's genotype contributes to this variability. Specifically, cytochrome P450 2D6 (CYP2D6) genotype has important relevance for response to opioid analgesics that depend on CYP2D6 for bioactivation. Poor metabolizers (PMs) have lower concentrations of active metabolites of codeine (morphine), tramadol (O-desmethyltramadol), oxycodone (oxymorphone), and hydrocodone (hydromorphone), compared to extensive metabolizers (EMs). Morphine and O-desmethyltramadol have 200-fold greater affinity for the µ-opioid receptor than the parent compound, whereas oxymorphone and hydromorphone have 40-fold and 10-fold higher receptor affinity compared to their parent compounds, respectively. Consequently, PMs may fail to derive pain relief from these opioids compared to EMs. Interestingly, the occurrence of side effects may not differ between PMs and EMs so that while PMs may get little to no pain relief from certain opioid analgesics, they may still experience troublesome adverse effects. Intermediate metabolizers (IMs) are also expected to have reduced analgesic response based on their significant reduction in enzyme activity. Conversely, individuals with the UM phenotype may have toxic concentrations of active opioid metabolites, with reports of life-threatening toxicity and death. The µ-opioid receptor gene (OPRM1) is the primary binding site for endogenous opioid peptides and opioid analgesics, and may have additional contributions to opioid response. The investigators propose to examine the effect of CYP2D6 genotype-guided pain management on cancer pain control in study participants and the additional effect of the OPRM1 genotype on response to opioids.

DETAILED DESCRIPTION:
This will be a randomized, open label, multi-site clinical trial conducted in UF Health Cancer Center in Gainesville, FL and in Moffitt Cancer Center in Tampa, FL. Each site will be responsible for overseeing patient care and research at their respective facility. This research will examine pain-related outcomes with CYP2D6-guided cancer pain management for study participants. In addition, the investigators will evaluate a prospective cohort study in the same population examining the effect of OPRM1 genetic variants on pain relief and adverse drug effects over time.

Participants will be randomized in a 1:1 manner to receive CYP2D6 genotype-guided (n=50) or non-genotype-guided (traditional, n=50) selection of pain medication. Patients in the genotype arm will be genotyped at baseline for CYP2D6 variants. Participants will fill out the the Brief Pain Inventory-Short Form (BPI-SF) and M.D. Anderson Symptom Inventory (MDASI) questionnaires at baseline. Then, during the clinical visits the same questionnaires will be done during weeks 2, 4, 6, and 8 or by telephone or electronic survey.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically or cytologically proven solid tumor with or without metastasis
* Receiving treatment at UF Health Cancer Center for outpatient pain management with an opioid

Exclusion Criteria:

* Undergone surgery within the last three months or are scheduled to undergo surgery during the study period (4 weeks)
* Documented psychiatric or neurological condition that would interfere with study participation
* Liver transplant
* Allergic to opioids

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2016-04; Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
Brief Pain Inventory-Short Form (BPI-SF) will be used to evaluate pain management and interference between the groups. | Change in baseline, weeks 2, 4, 6 and 8.
  Brief Pain Inventory-Short Form (BPI-SF) is a 9 item self-administered questionnaire used to evaluate the severity of a patient's pain and the impact of this pain on the patient's daily functioning. This is a 10-point scale with 0 being the best possible score, meaning "no pain", and 10 being the worst possible score, meaning "pain as bad as you can imagine".
MD Anderson Symptom Inventory (MDASI) will be used to evaluate symptom interference between the groups. | Change in baseline, weeks 2, 4, 6 and 8.
  MD Anderson Symptom Inventory (MDASI) modules augment the 19 core MDASI symptom and interference items with additional items identified as unique to a particular patient population. This is a 10-point scale with 0 being the best possible score, meaning "did not interfere" and 10 being the worst possible score, meaning "interfered completely".

SECONDARY OUTCOMES:
Observe Differences in Pain Control and Pain Interference between the number of participants based on OPRM1 Genotype | week 8
  At the end of the study, all participants will be genotyped for OPRM1 and evaluated for pain control (as assessed by the BPI-SF).
Observe Differences in Symptom Interference between the number of participants based on OPRM1 Genotype | week 8
  At the end of the study, all participants will be genotyped for OPRM1 and evaluated for symptom interference (as assessed by the MDASI).
Observe Differences in Opioid Doses between the number of participants based on OPRM1 Genotype | week 8
  At the end of the study, all participants will be genotyped for OPRM1 and evaluated for opioid dose (as assessed in morphine equivalent doses).

CONTACTS AND LOCATIONS:
Overall Officials: Larisa H Cavallari, PharmD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - University of Florida, Gainesville, Florida
  - H. Lee Moffitt Cancer Center & Research Institute, Tampa, Florida

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mosley SA, Cicali E, Del Cueto A, Portman DG, Donovan KA, Gong Y, Langaee T, Gopalan P, Schmit J, Starr JS, Silver N, Chang YD, Rajasekhara S, Smith JE, Soares HP, Clare-Salzler M, Starostik P, George TJ, McLeod HL, Fillingim RB, Hicks JK, Cavallari LH. CYP2D6-guided opioid therapy for adults with cancer pain: A randomized implementation clinical trial. Pharmacotherapy. 2023 Dec;43(12):1286-1296. doi: 10.1002/phar.2875. Epub 2023 Sep 21. PMID 37698371
- [Derived] Mosley SA, Hicks JK, Portman DG, Donovan KA, Gopalan P, Schmit J, Starr J, Silver N, Gong Y, Langaee T, Clare-Salzler M, Starostik P, Chang YD, Rajasekhara S, Smith JE, Soares HP, George TJ Jr, McLeod HL, Cavallari LH. Design and rational for the precision medicine guided treatment for cancer pain pragmatic clinical trial. Contemp Clin Trials. 2018 May;68:7-13. doi: 10.1016/j.cct.2018.03.001. Epub 2018 Mar 10. PMID 29535047